CLINICAL TRIAL: NCT04171947
Title: Medical Device Matuzalem Flavonoid Tea Extract Vaginal Ovule for the Correction of the Imbalance in the Vaginal Environment- Prospective, Multicentric, Two-arm, Randomized, Vehicle-controlled, Blinded, Comparative Clinical Trial
Brief Title: Vaginal Ovule With Flavonoid Tea Extract for the Correction of Imbalance in the Vaginal Environment
Acronym: MAT072017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Value Outcomes Ltd. (Other)
Collaborators: Matuzalem.com-cz, s.r.o. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAT072017
Record Dates: First submitted 2019-11-13; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Vaginosis, Bacterial; Vaginal Flora Imbalance
Keywords: Tea; Polyphenols; Nugent score; Antioxidants; Vaginal pH; complementary medicine
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Intervention Model Description: vehicle-controlled two-arm
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: blinded from the perspective of the participant, investigator, laboratory analyst and data analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Matuzalem (Experimental): Tea extract vaginal ovule daily for 7 consecutive days
  Interventions: Device: Matuzalem ovule
- Vehicle (Sham Comparator): Polyethylene glycol vaginal ovule daily for 7 consecutive days
  Interventions: Device: Vehicle ovule

INTERVENTIONS:
Device: Matuzalem ovule — vaginal ovule with 2 mg tea extract
  Arms: Matuzalem
Device: Vehicle ovule — polyethylene glycol vaginal ovule
  Arms: Vehicle

SUMMARY:
Randomized, blinded vehicle-controlled multicenter clinical trial (MAT072017) to determine the effect of vaginal ovules containing 2 mg of the tea extract Matuzalem on the subjective symptoms (5-point scale pruritus (itching), dolor (pain), rubor (redness), fluor (discharge), and fetor (odor)), and objective symptoms (pH, Nugent score) of bacterial vaginosis. An ovule containing only the vehicle (polyethylene glycol 3000 S) was used as a control. The study was blinded from the perspective of the subject, investigator, laboratory personnel and data analyst.

DETAILED DESCRIPTION:
The objective was to determine whether vaginal ovule with tea extract once-daily for 5-7 days improves symptoms of intermediate vaginal flora and prevents the development of bacterial vaginosis.

Composite primary endpoint designed as a drop in the Nugent score, vaginal pH, or improvement of subjective symptoms was compared between the active and vehicle (polyethylene-glycol) arm after 7 days of application and following 7 days after the application.

Secondary outcome measures were (1) Correction of the vaginal environment (as previously defined) 7 days after the completion of the prescribed 7-day regimen (day 14); (2) change in each parameter separately; (3) change in individual subjective symptoms, (4) exploratory analysis of the microbial environment at each subject visit.

The study was approved and supervised by the National authority and Ethics committee and prospectively registered in the Czech national medical device trial registry RZPRO and the European medical device trial registry EUDAMED.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal participants
* disturbed vaginal environment
* not in need of antibiotic or antimycotic treatment
* participants were citizens of the Czech Republic
* age between 18 and 55 years
* either a vaginal pH > 4.5 or/and vaginal discomfort
* able to follow the prescribed regimen
* informed consents prior to any intervention, including diagnostic procedures.

Exclusion Criteria:

* no vaginal bleeding of unknown aetiology
* hypersensitivity
* pregnancy
* lactation
* period during enrollment
* antibiotics in the previous 30 days
* treated with any products with similar indication
* acute urogenital infection
* diabetes mellitus
* advanced oncologic disease
* participant to other trial
* Nugent score above 6

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 274 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Composite endpoint (vaginal pH, Nugent score, subjective symptoms via questionnaire) after treatment completion | following 7 days of the ovule daily application
  Correction of the vaginal environment after 7 days of once-daily application of the ovule was defined as: a drop-in Nugent score to < 4 and/or a drop in vaginal pH to < 4.5, or a subjective improvement in at least 2 symptoms by at least 2 points on a 5-point scale in patients whose baseline pH was < 4.5 and NS < 4. Subjective symptoms: Pruritus, dolor, rubor, fluor and fetor reported by the patient on 5-point scale (0=no problem to 4=severe problem)

SECONDARY OUTCOMES:
Composite endpoint (vaginal pH, Nugent score, subjective symptoms via questionnaire) after 7 days since treatment completion | 7 days after the completion of the 7-day treatment
  Correction of the vaginal environment after 7 days after treatment completion defined as: a drop-in NS to < 4 and/or a drop in vaginal pH to < 4.5, or a subjective improvement in at least 2 symptoms by at least 2 points on a 5-point scale in patients whose baseline pH was < 4.5 and NS < 4. Subjective symptoms: Pruritus, dolor, rubor, fluor and fetor reported by the patient on 5-point scale (0=no problem to 4=severe problem)
Change in the pH alone after treatment completion | following 7 days of the ovule daily application
  Correction of the pH measured via pH strips
Change in the Nugent score alone after treatment completion | following 7 days of the ovule daily application
  Nugent score determined under 1000x magnification
Change in the subjective symptoms (questionnaire) after treatment completion | following 7 days of the ovule daily application
  Pruritus, dolor, rubor, fluor and fetor reported by the patient on 5-point scale (0=no problem to 4=severe problem)
Change in the pH alone after 7 days since treatment completion | 7 days after the completion of the 7-day treatment
  Correction of the pH measured via pH strips
Change in the Nugent score alone 7 days after treatment completion | 7 days after the completion of the 7-day treatment
  Nugent score determined under 1000x magnification
Change in the subjective symptoms (questionnaire) 7 days after treatment completion | 7 days after the completion of the 7-day treatment
  Pruritus, dolor, rubor, fluor and fetor reported by the patient on 5-point scale (0=no problem to 4=severe problem)
Exploratory analysis of the microbial environment after treatment completion: squamous epithelial cells | following 7 days of the ovule daily application
  Quantification of: squamous epithelial cells under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: squamous epithelial cells | 7 days after the completion of the 7-day treatment
  Quantification of: squamous epithelial cells under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: clue cells | following 7 days of the ovule daily application
  Quantification of clue cells under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: clue cells | 7 days after the completion of the 7-day treatment
  Quantification of clue cells under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: mixed flora | following 7 days of the ovule daily application
  Quantification of mixed flora under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: mixed flora | 7 days after the completion of the 7-day treatment
  Quantification of mixed flora under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: yeast as pseudomycelia | following 7 days of the ovule daily application
  Quantification of yeast as pseudomycelia under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: yeast as pseudomycelia | 7 days after the completion of the 7-day treatment
  Quantification of yeast as pseudomycelia under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: Gram negative diplococci | following 7 days of the ovule daily application
  Quantification of: Gram negative diplococci under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: Gram negative diplococci | 7 days after the completion of the 7-day treatment
  Quantification of: Gram negative diplococci under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: fibrous Lactobacillus | following 7 days of the ovule daily application
  Quantification of: fibrous Lactobacillus under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: fibrous Lactobacillus | 7 days after the completion of the 7-day treatment
  Quantification of: fibrous Lactobacillus under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: Gardnerella | following 7 days of the ovule daily application
  Quantification of: Gardnerella under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: Gardnerella | 7 days after the completion of the 7-day treatment
  Quantification of: Gardnerella under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: spirochetes | following 7 days of the ovule daily application
  Quantification of: spirochetes under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: spirochetes | 7 days after the completion of the 7-day treatment
  Quantification of: spirochetes under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: parabasal epithelial cells | following 7 days of the ovule daily application
  Quantification of: parabasal epithelial cells under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: parabasal epithelial cells | 7 days after the completion of the 7-day treatment
  Quantification of: parabasal epithelial cells under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: leukocytes | following 7 days of the ovule daily application
  Quantification of: leukocytes under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: leukocytes | 7 days after the completion of the 7-day treatment
  Quantification of: leukocytes under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: yeast as blastospores | following 7 days of the ovule daily application
  Quantification of: yeast as blastospores under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: yeast as blastospores | 7 days after the completion of the 7-day treatment
  Quantification of: yeast as blastospores under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: Gram pos. cocci in chains | following 7 days of the ovule daily application
  Quantification of: Gram pos. cocci in chains under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: Gram pos. cocci in chains | 7 days after the completion of the 7-day treatment
  Quantification of: Gram pos. cocci in chains under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: Lactobacillus | following 7 days of the ovule daily application
  Quantification of: Lactobacillus under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: Lactobacillus | 7 days after the completion of the 7-day treatment
  Quantification of: Lactobacillus under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: Mobilincus | following 7 days of the ovule daily application
  Quantification of: Mobilincus under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: Mobilincus | 7 days after the completion of the 7-day treatment
  Quantification of: Mobilincus under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: Leptotrichia | following 7 days of the ovule daily application
  Quantification of: Leptotrichia under 1000x magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: Leptotrichia | 7 days after the completion of the 7-day treatment
  Quantification of: Leptotrichia under 1000x magnification
Exploratory analysis of the microbial environment after treatment completion: Trichomonas vaginalis | following 7 days of the ovule daily application
  Quantification of: Trichomonas vaginalis under 1000 magnification
Exploratory analysis of the microbial environment after 7 days after treatment completion: Trichomonas vaginalis | 7 days after the completion of the 7-day treatment
  Quantification of: Trichomonas vaginalis under 1000 magnification

CONTACTS AND LOCATIONS:
Overall Officials: Tomáš Doležal, MD et PhD, Study Director — Value Outcomes Ltd.; Luboš Chadim, MVDr, Study Chair — Matuzalem.com-cz, s.r.o.
Locations (14):
- Czechia (14):
  - Centrum ambulantní gynekologie a primární péče, s.r.o., Brno, Czech Republic
  - MUDr. Milan Kučera. s.r.o., Kladno, Czech Republic
  - MUDr. Eva Novotná - FEMCARE s.r.o., Odolena Voda, Czech Republic
  - OB/GYN Associates, s.r.o., Prague, Czech Republic
  - MediStar s.r.o., Prague, Czech Republic
  - MUDr. Michal Jelšík, Prague, Czech Republic
  - Gyn Por Ivf MUDr. Samer Asad s.r.o., Prague, Czech Republic
  - Mediva s.r.o., Prague, Czech Republic
  - GYNEKOLOGIE Studentský dům s.r.o., Prague, Czech Republic
  - LEVRET s.r.o., Prague, Czech Republic
  - T.B. Gyn s.r.o., Prague, Czech Republic
  - Gynelav s.r.o., Prague, Czech Republic
  - GYNEDAN s.r.o., Prague, Czech Republic
  - MUDr.Tereza Šmrhová-Kovács, Tábor, Czech Republic

IPD SHARING:
Plan to Share IPD: No
Secondary analyses in progress